CLINICAL TRIAL: NCT02925234
Title: A Dutch National Study on Behalf of the CPCT to Facilitate Patient Access to Commercially Available, Targeted Anti-cancer Drugs to Determine the Potential Efficacy in Treatment of Advanced Cancers With a Known Molecular Profile
Brief Title: The Drug Rediscovery Protocol (DRUP Trial)
Acronym: DRUP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Amgen (Industry); AstraZeneca (Industry); Bayer (Industry); Bristol-Myers Squibb (Industry); Novartis (Industry); Roche Pharma AG (Industry); Merck Sharp & Dohme LLC (Industry); Boehringer Ingelheim (Industry); Ipsen (Industry); Eisai Inc. (Industry); Pfizer (Industry); Clovis Oncology - Pharma and (Unknown); Eli Lilly and Company (Industry); Janssen, LP (Industry); GlaxoSmithKline (Industry); Incyte Corporation (Industry); Dutch Cancer Society (Other); Stelvio for Life (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M15DRU
Record Dates: First submitted 2016-08-26; First posted 2016-10-05 (Estimated); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Cancer; Tumors; Neoplasm; Neoplasia
Keywords: Molecular tumor profile; Multidisciplinary tumor board; Antitumor drugs; Molecular Targeted Therapy; Drug Repositioning; Off-Label Use; Sequence Analysis, DNA
MeSH Terms: conditions — Neoplasms | interventions — Panitumumab; olaparib; dabrafenib; nilotinib; trametinib; Erlotinib Hydrochloride; Trastuzumab; pertuzumab; Vemurafenib; cobimetinib; HhAntag691; regorafenib; Nivolumab; Afatinib; ribociclib; lenvatinib; pembrolizumab; durvalumab; rucaparib; Axitinib; palbociclib; Crizotinib; Sunitinib; cabozantinib; abemaciclib; alectinib; atezolizumab; Bevacizumab; Ipilimumab; entrectinib; talazoparib; dacomitinib; lorlatinib; erdafitinib; Alpelisib; niraparib; pemigatinib; selpercatinib; tepotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (37):
- Panitumumab (Experimental): Panitumumab for patients with a molecular tumor profile that can potentially be targeted by Panitumumab.
  Interventions: Drug: Panitumumab
- Olaparib (Experimental): Olaparib for patients with a molecular tumor profile that can potentially be targeted by Olaparib.
  Interventions: Drug: Olaparib
- Dabrafenib (Experimental): Dabrafenib for patients with a molecular tumor profile that can potentially be targeted by Dabrafenib.
  Interventions: Drug: Dabrafenib
- Nilotinib (Experimental): Nilotinib for patients with a molecular tumor profile that can potentially be targeted by nilotinib.
  Interventions: Drug: Nilotinib
- Trametinib (Experimental): Trametinib for patients with a molecular tumor profile that can potentially be targeted by trametinib.
  Interventions: Drug: Trametinib
- Erlotinib (Experimental): Erlotinib for patients with a molecular tumor profile that can potentially be targeted by erlotinib.
  Interventions: Drug: Erlotinib
- Trastuzumab & Pertuzumab (combination) (Experimental): Trastuzumab and Pertuzumab (combination treatment) for patients with a molecular tumor profile that can potentially be targeted by Trastuzumab and Pertuzumab.
  Interventions: Drug: Trastuzumab and Pertuzumab (combination treatment)
- Vemurafenib & Cobimetinib (combination) (Experimental): Vemurafenib and Cobimetinib (combination treatment) for patients with a molecular tumor profile that can potentially be targeted by Vemurafenib and Cobimetinib.
  Interventions: Drug: Vemurafenib and Cobimetinib (combination treatment)
- Vismodegib (Experimental): Vismodegib for patients with a molecular tumor profile that can potentially be targeted by vismodegib.
  Interventions: Drug: Vismodegib
- Regorafenib (Experimental): Regorafenib for patients with a molecular tumor profile that can potentially be targeted by regorafenib.
  Interventions: Drug: Regorafenib
- Nivolumab (Experimental): Nivolumab for patients with a molecular tumor profile that can potentially be targeted by nivolumab.
  Interventions: Drug: Nivolumab
- Afatinib (Experimental): Afatinib for patients with a molecular tumor profile that can potentially be targeted by Afatinib.
  Interventions: Drug: Afatinib
- Dabrafenib & trametinib (combination) (Experimental): Dabrafenib and trametinib (combination treatment) for patients with a molecular tumor profile that can potentially be targeted by Dabrafenib and trametinib.
  Interventions: Drug: Dabrafenib and trametinib
- Ribociclib (Experimental): Ribociclib for patients with a molecular tumor profile that can potentially be targeted by Ribociclib.
  Interventions: Drug: Ribociclib
- Lenvatinib (Experimental): Lenvatinib for patients with a molecular tumor profile that can potentially be targeted by Lenvatinib.
  Interventions: Drug: Lenvatinib
- Pembrolizumab (Experimental): Pembrolizumab for patients with a molecular tumor profile that can potentially be targeted by Pembrolizumab.
  Interventions: Drug: Pembrolizumab
- Durvalumab (Experimental): Durvalumab for patients with a molecular tumor profile that can potentially be targeted by Durvalumab.
  Interventions: Drug: Durvalumab
- Rucaparib (Experimental): Rucaparib for patients with a molecular tumor profile that can potentially be targeted by Rucaparib.
  Interventions: Drug: Rucaparib
- Axitinib (Experimental): Axitinib for patients with a molecular tumor profile that can potentially be targeted by Axitinib.
  Interventions: Drug: Axitinib
- Palbociclib (Experimental): Palbociclib for patients with a molecular tumor profile that can potentially be targeted by Palbociclib.
  Interventions: Drug: Palbociclib
- Crizotinib (Experimental): Crizotinib for patients with a molecular tumor profile that can potentially be targeted by Crizotinib.
  Interventions: Drug: Crizotinib
- Sunitinib (Experimental): Sunitinib for patients with a molecular tumor profile that can potentially be targeted by Sunitinib.
  Interventions: Drug: Sunitinib
- Cabozantinib (Experimental): Cabozantinib for patients with a molecular tumor profile that can potentially be targeted by Cabozantinib.
  Interventions: Drug: Cabozantinib
- Abemaciclib (Experimental): Abemaciclib for patients with a molecular tumor profile that can potentially be targeted by Abemaciclib.
  Interventions: Drug: Abemaciclib
- Alectinib (Experimental): Alectinib for patients with a molecular tumor profile that can potentially be targeted by Alectinib.
  Interventions: Drug: Alectinib
- Atezolizumab/bevacizumab (Experimental): Atezolizumab and bevacizumab (combination treatment) for patients with a molecular tumor profile that can potentially be targeted by Atezolizumab and bevacizumab.
  Interventions: Drug: Atezolizumab and Bevacizumab
- Ipilimumab/nivolumab (Experimental): Ipilimumab and nivolumab (combination treatment) for patients with a molecular tumor profile that can potentially be targeted by Ipilimumab and nivolumab.
  Interventions: Drug: Ipilimumab and nivolumab
- Entrectinib (Experimental): Entrectinib for patients with a molecular tumor profile that can potentially be targeted by entrectinib.
  Interventions: Drug: Entrectinib
- Talazoparib (Experimental): Talazoparib for patients with a molecular tumor profile that can potentially be targeted by talazoparib.
  Interventions: Drug: Talazoparib
- dacomitinib (Experimental): Dacomitinib for patients with a molecular tumor profile that can potentially be targeted by dacomitinib.
  Interventions: Drug: Dacomitinib
- Lorlatinib (Experimental): Lorlatinib for patients with a molecular tumor profile that can potentially be targeted by lorlatinib.
  Interventions: Drug: Lorlatinib
- Erdafitinib (Experimental): Erdafitinib for patients with a molecular tumor profile that can potentially be targeted by erdafitinib.
  Interventions: Drug: Erdafitinib
- Alpelisib (Experimental): Alpelisib for patients with a molecular tumor profile that can potentially be targeted by alpelisib.
  Interventions: Drug: Alpelisib
- Niraparib (Experimental): Niraparib for patients with a molecular tumor profile that can potentially be targeted by niraparib.
  Interventions: Drug: Niraparib
- Pemigatinib (Experimental): Pemigatinib for patients with a molecular tumor profile that can potentially be targeted by pemigatinib.
  Interventions: Drug: Pemigatinib
- Selpercatinib (Experimental): Selpercatinib for patients with a molecular tumor profile that can potentially be targeted by selpercatinib.
  Interventions: Drug: Selpercatinib
- Tepotinib (Experimental): Tepotinib for patients with a molecular tumor profile that can potentially be targeted by tepotinib.
  Interventions: Drug: Tepotinib

INTERVENTIONS:
Drug: Panitumumab — Panitumumab treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of panitumumab might be expected based on their molecular tumor profile.
  Other Names: Vectibix
  Arms: Panitumumab
Drug: Olaparib — Olaparib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of olaparib might be expected based on their molecular tumor profile.
  Other Names: Lynparza
  Arms: Olaparib
Drug: Dabrafenib — Dabrafenib treatment for patients with an mutated advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of dabrafenib might be expected based on their molecular tumor profile.
  Other Names: Tafinlar
  Arms: Dabrafenib
Drug: Nilotinib — Nilotinib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of nilotinib might be expected based on their molecular tumor profile.
  Other Names: Tasigna
  Arms: Nilotinib
Drug: Trametinib — Trametinib treatment for patients with an mutated advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of trametinib might be expected based on their molecular tumor profile.
  Other Names: Mekinist
  Arms: Trametinib
Drug: Erlotinib — Erlotinib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of erlotinib might be expected based on their molecular tumor profile.
  Other Names: Tarceva
  Arms: Erlotinib
Drug: Trastuzumab and Pertuzumab (combination treatment) — Trastuzumab and Pertuzumab treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of trastuzumab + pertuzumab might be expected based on their molecular tumor profile.
  Other Names: Herceptin + Perjeta
  Arms: Trastuzumab & Pertuzumab (combination)
Drug: Vemurafenib and Cobimetinib (combination treatment) — Vemurafenib + Cobimetinib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of Vemurafenib + Cobimetinib might be expected based on their molecular tumor profile.
  Other Names: Zelboraf + Cotellic
  Arms: Vemurafenib & Cobimetinib (combination)
Drug: Vismodegib — Vismodegib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of vismodegib might be expected based on their molecular tumor profile.
  Other Names: Erivedge
  Arms: Vismodegib
Drug: Regorafenib — Regorafenib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of vismodegib might be expected based on their molecular tumor profile.
  Other Names: Stivarga
  Arms: Regorafenib
Drug: Nivolumab — Nivolumab treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of nivolumab might be expected based on their molecular tumor profile.
  Other Names: Opdivo
  Arms: Nivolumab
Drug: Afatinib — Afatinib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of Afatinib might be expected based on their molecular tumor profile.
  Other Names: Giotrif
  Arms: Afatinib
Drug: Dabrafenib and trametinib — Dabrafenib + trametinib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of Dabrafenib + Trametinib might be expected based on their molecular tumor profile.
  Other Names: Tafinlar and Mekinist
  Arms: Dabrafenib & trametinib (combination)
Drug: Ribociclib — Ribociclib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of Ribociclib might be expected based on their molecular tumor profile.
  Other Names: Kisqali
  Arms: Ribociclib
Drug: Lenvatinib — Lenvatinib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of Lenvatinib might be expected based on their molecular tumor profile.
  Other Names: Lenvima
  Arms: Lenvatinib
Drug: Pembrolizumab — Pembrolizumab treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of Pembrolizumab might be expected based on their molecular tumor profile.
  Other Names: Keytruda
  Arms: Pembrolizumab
Drug: Durvalumab — Durvalumab treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of Durvalumab might be expected based on their molecular tumor profile.
  Other Names: MEDI4736
  Arms: Durvalumab
Drug: Rucaparib — Rucaparib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of Rucaparib might be expected based on their molecular tumor profile.
  Other Names: Rubraca
  Arms: Rucaparib
Drug: Axitinib — Axitinib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of Axitinib might be expected based on their molecular tumor profile.
  Other Names: Inlyta
  Arms: Axitinib
Drug: Palbociclib — Palbociclib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of Palbociclib might be expected based on their molecular tumor profile.
  Other Names: Ibrance
  Arms: Palbociclib
Drug: Crizotinib — Crizotinib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of Crizotinib might be expected based on their molecular tumor profile.
  Other Names: Xalkori
  Arms: Crizotinib
Drug: Sunitinib — Sunitinib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of Sunitinib might be expected based on their molecular tumor profile.
  Other Names: Sutent
  Arms: Sunitinib
Drug: Cabozantinib — Cabozantinib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of Cabozantinib might be expected based on their molecular tumor profile.
  Other Names: Cabometyx
  Arms: Cabozantinib
Drug: Abemaciclib — Abemaciclib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of Abemaciclib might be expected based on their molecular tumor profile.
  Other Names: Verzenios
  Arms: Abemaciclib
Drug: Alectinib — Alectinib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of Alectinib might be expected based on their molecular tumor profile.
  Other Names: Alecensa
  Arms: Alectinib
Drug: Atezolizumab and Bevacizumab — Atezolizumab + Bevacizumab treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of Atezolizumab + Bevacizumab might be expected based on their molecular tumor profile.
  Other Names: Tecentriq and Avastin
  Arms: Atezolizumab/bevacizumab
Drug: Ipilimumab and nivolumab — Ipilimumab+nivolumab treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of ipilimimab + nivolumab might be expected based on their molecular tumor profile.
  Other Names: Yervoy and Opdivo
  Arms: Ipilimumab/nivolumab
Drug: Entrectinib — Entrectinib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of entrectinib might be expected based on their molecular tumor profile.
  Other Names: Rozlytrek
  Arms: Entrectinib
Drug: Talazoparib — Talazoparib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of talazoparib might be expected based on their molecular tumor profile.
  Other Names: Talzenna
  Arms: Talazoparib
Drug: Dacomitinib — Dacomitinib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of dacomitinib might be expected based on their molecular tumor profile.
  Other Names: Vizimpro
  Arms: dacomitinib
Drug: Lorlatinib — Lorlatinib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of lorlatinib might be expected based on their molecular tumor profile.
  Other Names: Lorviqua
  Arms: Lorlatinib
Drug: Erdafitinib — Erdafitinib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of erdafitinib might be expected based on their molecular tumor profile.
  Other Names: Balversa
  Arms: Erdafitinib
Drug: Alpelisib — Alpelisib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of alpelisib might be expected based on their molecular tumor profile.
  Other Names: Piqray
  Arms: Alpelisib
Drug: Niraparib — Niraparib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of niraparib might be expected based on their molecular tumor profile.
  Other Names: Zejula
  Arms: Niraparib
Drug: Pemigatinib — Pemigatinib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of pemigatinib might be expected based on their molecular tumor profile.
  Other Names: Pemazyre
  Arms: Pemigatinib
Drug: Selpercatinib — Selpercatinib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of selpercatinib might be expected based on their molecular tumor profile.
  Other Names: Retsevmo
  Arms: Selpercatinib
Drug: Tepotinib — Tepotinib treatment for patients with an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma, who are not eligible for on-label treatment but for whom anti-tumor activity of tepotinib might be expected based on their molecular tumor profile.
  Other Names: Tepmetko
  Arms: Tepotinib

SUMMARY:
This is a prospective, non-randomized clinical trial that aims to describe the efficacy and toxicity of commercially available, targeted anticancer drugs* prescribed for treatment of patients with advanced cancer with a potentially actionable variant as revealed by a genomic or protein expression test. The study also aims to simplify patient access to approved targeted therapies that are contributed to the program by collaborating pharmaceutical companies and to perform next generation sequencing on tumor biopsies for biomarker analyses. Eligible patients have an advanced solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma for which standard treatment options are no longer available and acceptable performance status and organ function. A genomic or protein expression test must have been performed on the tumor and the results must identify at least one potentially actionable molecular variant as defined in the protocol. Results from the molecular profiling test will be used to determine an appropriate drug(s) from among those available in the protocol. The choice of drug will be supported by a list of potential profiles, a molecular tumor board, a knowledge library and by study coordinators for review and approval of the match. The protocol-specified treatment will be administered to the patient once any drug-specific eligibility criteria are confirmed and a fresh pre-treatment biopsy is performed for future genetic studies. All patients who receive treatment with a drug available in the protocol will be followed for standard efficacy outcomes including tumor response, progression-free and overall survival as well as duration of treatment. In addition, treatment related toxicity will be evaluated.

DETAILED DESCRIPTION:
Problem description: evidence is building that matching targeted agents to tumor characteristics can improve outcomes. Such reports have fueled interest among patients and physicians to use molecular testing for treatment planning when standard treatment options have been exhausted. When oncologists aim to provide such personalized treatment to their patients though, obtaining the drugs can be challenging since off-label prescribing, while legal, is generally not reimbursed by insurance companies. Furthermore, outcomes of off-label treatment in routine clinical practice are not systematically recorded. As a result, the research and clinical communities have limited insight in these outcomes, leading to repetitive use of ineffective treatment for some tumor types, while effective treatment strategies might be missed for others. The latter is especially relevant for 'orphan diseases', that are too rare to conduct formal phase II and III trials. In summary, there is a lack of access to potentially effective therapy on one hand, and a lack of knowledge on broader use of such therapies on the other, altogether leading to sub-optimal use of available resources.

Envisioned solution and study aim: creation of a drug-access program, in which patients are treated with registered targeted therapy matched to their molecular tumor profile, and in which the outcomes of such therapies are recorded systematically, per tumor profile and tumor type (this is important since it is becoming increasingly clear that the tissue of origin is an important determinant of outcome of genetic abnormalities). We hereby aim to improve and broaden the use of registered targeted therapy, whilst facilitating patient access to such therapy.

Plan of investigation: patients will be treated with approved targeted agents, selected based on results of a molecular profiling test of the patient's tumor. Eligible patients will have exhausted standard treatment options, and their tumor must harbor a potentially actionable molecular variant as defined in the protocol. The study will provide a tumor board to help physicians understand the profiling test results and treatment options, and will enable insights about the utility of this approach. In addition, next generation sequencing will be performed on fresh tumor biopsies for additional biomarker discovery. Patients from the Netherlands and the USA will be included in two similar though independent protocols (DRUP and TAPUR), allowing data-exchange and empowering of both trials.

Expected outcome: early signs of clinical activity of approved drugs outside their label, providing effective personalized treatment options, improved patient outcomes and access to targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age >18 years) patient with a histologically-proven locally advanced or metastatic solid tumor, multiple myeloma or B cell non-Hodgkin lymphomawith symptomatic disease progression or progression according to RECIST-criteria after standard anti-cancer treatment or for whom no such treatment is available or indicated.

   * For patients with a primary brain tumor: Histologically confirmed recurrent or de novo primary brain tumor, with unequivocal progression after prior therapy, at least 3 months after radiotherapy (either first line chemo-radiotherapy or re-irradiation), and with stable or decreasing dosage of steroids for at least 7 days prior to the baseline MRI scan.
2. ECOG performance status 0-2
3. Patients must have acceptable organ function as defined below. However, specific inclusion/exclusion criteria specified in the drug-specific study manual will take precedence:

   1. Absolute neutrophil count ≥ 1.5 x 109/l
   2. Hemoglobin > 5.6 mmol/l
   3. Platelets > 75 x 109/l
   4. Total bilirubin < 2 x ULN
   5. AST (SGOT) and ALT (SGPT) < 2.5 x institutional ULN (or < 5 x ULN in patients with known hepatic metastases)
   6. Serum creatinine ≤ 1.5 × ULN or calculated or measured creatinine clearance ≥ 50 mL/min/1.73 m2
4. Patients must have objectively measurable disease (by physical or radiographic examination, according to RECIST v1.1 for patients with solid tumors, or according to IMWG, Lugano, RANO or GCIG criteria, resp., for patients with multiple myeloma, non-Hodgkin lymphoma, glioblastoma or ovarian cancer in case of CA125-based evaluation (please refer to appendices for further details).
5. Results must be available from a tumor genomic or protein expression test. Eligible tests may include any of the following technologies: fluorescence in situ hybridization (FISH), polymerase chain reaction (PCR), comparative genomic hybridization (CGH), next generation sequencing (NGS) or immunohistochemistry (IHC). The test may have been performed on the primary tumor or a metastatic deposit, in a diagnostic laboratory or within the context of another CPCT study, and must reveal a potentially actionable variant as defined in Section 5. The test results (full pathology or molecular diagnostics report) must be uploaded in the eCRF.
6. Patients must have a tumor profile for which treatment with one of the FDA and / or EMA approved (or under revision for approval) targeted anti-cancer drugs included in this study has potential clinical benefit based on preclinical data or clinical information (see section 5).
7. new (obtained ≤2 months before inclusion, and without any type of anti-cancer therapy within those ≤2 months) fresh frozen tumor biopsy specimen for extensive biomarker testing is mandatory before the start of treatment with a targeted agent included in the protocol. Alternatively, fresh frozen tumor tissue acquired in the context of a standard care procedure may be used, provided that no systemic anti-cancer treatment was given between the procedure and start of study treatment within DRUP.

   The following exceptions are made:

   a. An exception is made for patients with a primary brain tumor, only if the mandatory DRUP pre-treatment biopsy for biomarker analysis cannot safely be obtained:
   1. The fresh frozen tumor biopsy sample may be replaced by fresh frozen tumor tissue, obtained earlier from recurrent disease, as part of standard of care surgical procedure (i.e., performed at progression)
   2. If no fresh frozen tumor tissue is available for NGS, and the risk of obtaining a new tumor biopsy is considered too high, no biopsy will be required. In this case, the study coordinators must be informed in advance, and there will be no reimbursement for the biopsy procedure.

   b. In case WGS is performed on tumor tissue outside the context of a clinical trial before inclusion, and without any type of anti-cancer therapy between the collection of tissue and inclusion in DRUP, this can replace the DRUP pre-treatment biopsy, provided that the patient gives consent to use his/her WGS data for biomarker analysis in DRUP.

   c. An exception is made for patients that underwent an allogeneic hematopoietic stem cell transplantation prior to study enrollment, since this will prevent a correct WGS analysis due to a mismatch between the biopsy specimen and the required blood sample.
8. Ability to understand and the willingness to sign a written informed consent document.
9. For orally administered drugs, the patient must be able to swallow and tolerate oral medication and must have no known malabsorption syndrome.
10. Because of the risks of drug treatment to the developing foetus, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation, and for four months following completion of study therapy. Male patients should avoid impregnating a female partner. Male patients, even if surgically sterilized, (i.e. post-vasectomy) must agree to one of the following: practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug, or completely abstain from sexual intercourse.

Exclusion Criteria:

1. Ongoing toxicity > grade 2, other than alopecia.
2. Patient is receiving any other anti-cancer therapy (cytotoxic, biologic, radiation, or hormonal other than for replacement). Required wash out period prior to starting study treatment is at least two weeks. An exception is made for:

   * Patients suffering from CRPC are allowed to continue androgen deprivation therapy.
   * Medications that are prescribed for supportive care but may potentially have an anti-cancer effect (e.g., megestrol acetate, bisphosphonates). These medications must have been started ≥ 1 week prior to enrollment on this study.
3. Patient is pregnant or nursing.
4. Patients with known active progressive brain metastases. Patients with previously treated brain metastases are eligible, provided that the patient has not experienced a seizure or had a clinically significant change in neurological status within the 3 months prior to registration. All patients with previously treated brain metastases must be stable for at least 1 month after completion of treatment and off steroid treatment prior to study enrollment.

   * Additional exclusion criteria specific for glioblastoma patients:
   1. Patients who require anti-convulsant therapy must be taking non-enzyme inducing antiepileptic drugs (non-EIAED). EIAED are prohibited. Patients previously on EIAED must be switched to non-EIAED at least 2 weeks prior to randomization.
   2. No radiotherapy within the three months prior to the diagnosis of progression.
   3. No radiotherapy with a dose over 65 Gy, stereotactic radiosurgery or brachytherapy unless the recurrence is histologically proven.
5. Patients with clinically significant preexisting cardiac conditions, including uncontrolled or symptomatic angina, uncontrolled atrial or ventricular arrhythmias, or symptomatic congestive heart failure are not eligible.
6. Patients with known left ventricular ejection fraction (LVEF) < 40% are not eligible
7. Patients with stroke (including TIA) or acute myocardial infarction within 3 months before the first dose of study treatment are not eligible
8. Patients with any other clinically significant medical condition which, in the opinion of the treating physician, makes it undesirable for the patient to participate in the study or which could jeopardize compliance with study requirements including, but not limited to: ongoing or active infection, significant uncontrolled hypertension, or severe psychiatric illness/social situations.

For each drug included in this protocol, specific inclusion and exclusion criteria (based on the Package Insert or manufacturers recommendations) may also apply. These can be found in the supplemental information about each agent included in the drug-specific study manuals. Drug-specific inclusion and exclusion criteria will take precedence over the inclusion/exclusion criteria listed above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1550 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients that are treated based on their molecular tumor profile | 6 months after treatment initiation (estimated average)
  Primary outcome measure 1 is the percentage of submitted patients, that can be treated based on their molecular tumor profile within the context of this protocol.
Objective tumor response | 6 months after treatment initiation (estimated average)
  Primary outcome measure 2 is the proportion of study participants with an objective tumor response upon study treatment..
Stable disease | 6 months after treatment initiation (estimated average)
  Primary outcome measure 3 is the proportion of study participants that has stable disease (SD) during study treatment.
Treatment-related grade≥3 and serious adverse events | 6 months after treatment initiation (estimated average)
  Primary outcome measure 4 is the proportion of patients that experience treatment-related grade≥3 and /or serious adverse events.

SECONDARY OUTCOMES:
Progression-free survival | Up to 1 year after study completion
Overall survival | Up to 1 year after study completion
Duration of treatment on study (time on drug) | 6 months after treatment initiation (estimated average)

OTHER OUTCOMES:
Concordance between pre-treatment and historic mutational tumor profile | 2 months after treatment initiation (estimated average)
  Sequencing results of fresh pre-treatment biopsies will be available within 2 months after treatment initiation.

CONTACTS AND LOCATIONS:
Overall Officials: E.E. Voest, prof., Principal Investigator — The Netherlands Cancer Institute
Locations (36):
- Netherlands (36):
  - Noordwest ziekenhuisgroep Alkmaar (NWZ), Alkmaar
  - Ziekenhuisgroep Twente, Almelo
  - Meander medisch centrum, Amersfoort
  - Netherlands Cancer Institute, Amsterdam
  - Amsterdam UMC, locatie VUmc, Amsterdam
  - Amsterdam UMC, locatie AMC, Amsterdam
  - Onze Lieve Vrouwe Gasthuis (OLVG), Amsterdam
  - Gelre ziekenhuizen, Apeldoorn
  - Rijnstate ziekenhuis, Arnhem
  - Amphia Ziekenhuis, Breda
  - Reiner de Graaf Gasthuis, Delft
  - Deventer ziekenhuis, Deventer
  - Nij Smellinghe Ziekenhuis, Drachten
  - Ziekenhuis Gelderse Vallei, Ede
  - Maxima Medisch Centrum, Eindhoven
  - Zuyderland medisch centrum, Geleen
  - Rivas zorggroep, Gorinchem
  - Martini ziekenhuis, Groningen
  - University Medical Center Groningen, Groningen
  - Spaarne gasthuis, Haarlem
  - Tergooi MC, Hilversum
  - Treant zorggroep, Hoogeveen
  - Medisch Centrum Leeuwaarden, Leeuwarden
  - Leiden University Medical Center, Leiden
  - Maastricht University Medical Center, Maastricht
  - St. Antonius ziekenhuis, Nieuwegein
  - Radboud umc, Nijmegen
  - Bravis ziekenhuis, Roosendaal
  - St. Fransicus Gasthuis, Rotterdam
  - Erasmus MC, Rotterdam
  - Haaglanden medisch centrum, The Hague
  - Haga ziekenhuis, The Hague
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg
  - University Medical Center Utrecht, Utrecht
  - VieCuri medisch centrum, Venlo
  - Isala klinieken, Zwolle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Geurts BS, Zeverijn LJ, Leek LVM, van Berge Henegouwen JM, Hoes LR, van der Wijngaart H, van der Noort V, van de Haar J, van Ommen-Nijhof A, Kok M, Roepman P, Jansen AML, de Leng WWJ, de Jonge MJA, Hoeben A, van Herpen CML, Westgeest HM, Wessels LFA, Verheul HMW, Gelderblom H, Voest EE. Efficacy of Pembrolizumab and Biomarker Analysis in Patients with WGS-Based Intermediate to High Tumor Mutational Load: Results from the Drug Rediscovery Protocol. Clin Cancer Res. 2024 Sep 3;30(17):3735-3746. doi: 10.1158/1078-0432.CCR-24-0011. PMID 38630551
- [Derived] Zeverijn LJ, Looze EJ, Thavaneswaran S, van Berge Henegouwen JM, Simes RJ, Hoes LR, Sjoquist KM, van der Wijngaart H, Sebastian L, Geurts BS, Lee CK, de Wit GF, Espinoza D, Roepman P, Lin FP, Jansen AML, de Leng WWJ, van der Noort V, Leek LVM, de Vos FYFL, van Herpen CML, Gelderblom H, Verheul HMW, Thomas DM, Voest EE. Limited clinical activity of palbociclib and ribociclib monotherapy in advanced cancers with cyclin D-CDK4/6 pathway alterations in the Dutch DRUP and Australian MoST trials. Int J Cancer. 2023 Oct 1;153(7):1413-1422. doi: 10.1002/ijc.34649. Epub 2023 Jul 10. PMID 37424386
- [Derived] Geurts BS, Battaglia TW, van Berge Henegouwen JM, Zeverijn LJ, de Wit GF, Hoes LR, van der Wijngaart H, van der Noort V, Roepman P, de Leng WWJ, Jansen AML, Opdam FL, de Jonge MJA, Cirkel GA, Labots M, Hoeben A, Kerver ED, Bins AD, Erdkamp FGL, van Rooijen JM, Houtsma D, Hendriks MP, de Groot JB, Verheul HMW, Gelderblom H, Voest EE. Efficacy, safety and biomarker analysis of durvalumab in patients with mismatch-repair deficient or microsatellite instability-high solid tumours. BMC Cancer. 2023 Mar 4;23(1):205. doi: 10.1186/s12885-023-10663-2. PMID 36870947
- [Derived] van Berge Henegouwen JM, van der Wijngaart H, Zeverijn LJ, Hoes LR, Meertens M, Huitema ADR, Devriese LA, Labots M, Verheul HMW, Voest EE, Gelderblom H. Efficacy and toxicity of vemurafenib and cobimetinib in relation to plasma concentrations, after administration via feeding tube in patients with BRAF-mutated thyroid cancer: a case series and review of literature. Cancer Chemother Pharmacol. 2022 Jul;90(1):97-104. doi: 10.1007/s00280-022-04437-z. Epub 2022 May 22. PMID 35598186
- [Derived] Nakauma-Gonzalez JA, Rijnders M, van Riet J, van der Heijden MS, Voortman J, Cuppen E, Mehra N, van Wilpe S, Oosting SF, Rijstenberg LL, Westgeest HM, Zwarthoff EC, de Wit R, van der Veldt AAM, van de Werken HJG, Lolkema MPJ, Boormans JL. Comprehensive Molecular Characterization Reveals Genomic and Transcriptomic Subtypes of Metastatic Urothelial Carcinoma. Eur Urol. 2022 Apr;81(4):331-336. doi: 10.1016/j.eururo.2022.01.026. Epub 2022 Jan 25. PMID 35086719